CLINICAL TRIAL: NCT01644877
Title: A Phase II, Randomized, Double-blind, Placebo-controlled Study to Examine the Effects of DAS181 in Immunocompromised Subjects With Lower Respiratory Tract Parainfluenza Infection on Supplemental Oxygen
Acronym: DAS181-2-05
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ansun Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAS181-2-05
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Parainfluenza
MeSH Terms: conditions — Paramyxoviridae Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DAS181 (Experimental): DAS181-F02, 4.5 mg qd x 10 days
  Interventions: Drug: DAS181 dry powder, formulation F02
- Lactose Placebo (Placebo Comparator): placebo, 4.5 mg qd x 10 days
  Interventions: Drug: Lactose Placebo

INTERVENTIONS:
Drug: DAS181 dry powder, formulation F02
  Arms: DAS181
Drug: Lactose Placebo
  Arms: Lactose Placebo

SUMMARY:
This protocol will seek to enroll immunocompromised patients who are on supplemental oxygen and diagnosed with a parainfluenza infection.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥12 years
* Able to provide informed consent, child assent with parental consent or surrogate consent when applicable
* Currently on invasive mechanical ventilation or noninvasive positive pressure ventilation (CPAP or bilevel positive airway pressure) or requiring > 2LPM supplemental oxygen therapy to maintain O2 saturation > 90% due to hypoxemia
* Immunocompromised, as defined by one of the following: Autologous or Allogeneic hematopoietic cell transplantation (HSCT); Lung or lung-heart transplantation; Subjects treated with chemotherapy for hematologic malignancies; Subjects treated with chemotherapy for solid tumor malignancies
* Confirmed parainfluenza at screening by one of the following methods using any sample type: Respiratory Virus Panel, Direct fluorescent antibody (DFA), Qualitative/quantitative RT-PCR test for parainfluenza virus performed at the local laboratory (a confirmatory PCR test will be done at the central lab but is not required to start the patient on study).
* Confirmed PIV lower tract disease for subjects on mechanical ventilation will be defined as PIV detection in bronchoalveolar lavage (BAL) or biopsy within last 7 days of screening
* Confirmed PIV lower tract disease for subjects on non-invasive positive pressure ventilation or supplemental oxygen will be defined as all of the following within the last 7 days of screening: New pulmonary infiltrate on chest imaging and at least one PIV sign and/or symptom as defined in section 10.3.6
* Female subjects of child-bearing potential who are capable of conception must be post-menopausal (one year or greater without menses), surgically incapable of childbearing, or practicing two effective methods of birth control. Acceptable methods include abstinence, intrauterine device, spermicide, barrier, male partner surgical sterilization and hormonal contraception. A female subject ≥18 years of age and of child bearing potential must agree to practice two acceptable methods of birth control during the study period. All reproductive female subjects must have a negative serum pregnancy test during the screening visit.
* Male subjects must agree to use medically accepted form of contraception during the study period. Abstinence is an acceptable method of contraception.

Exclusion Criteria:

* Psychiatric or cognitive illness or recreational drug/alcohol use that, in the opinion of the principal investigator, would affect patient safety and/or compliance.
* Any significant finding in the patient's medical history or physical examination that, in the opinion of the investigator, would affect patient safety or compliance with the dosing schedule.
* In the opinion of the Investigator, subjects with a low chance of survival during the first 5 days of treatment.
* Subjects treated with oral, aerosolized or intravenous (IV) ribavirin for the treatment of PIV. A forty-eight hour (48 hr) wash out period prior to randomization is allowed.
* Subjects with a history of RSV or MPV
* Subjects taking any other investigational drug used to research or treat PIV.
* Subjects with a history of allergic reactions to lactose.
* Subjects with a history of documented Pseudomonas aeruginosa pneumonia confirmed radiographically and by culture from BAL.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2014-03; Primary Completion 2016-12-15 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
Clinical Stability | 45 days
  Clinical stability survival (CSS) rate is defined as subjects who meet the clinical stability criteria and are alive at Study Day 45 (Responders) compared to those who have not met clinical stability criteria or have expired regardless of stability status (Non-responders)

SECONDARY OUTCOMES:
Clinical Stability | 45 days
  Clinical stability (CS) rate excluding survival status: Clinical stability (CS) rate is defined as subjects who reached clinical stability criteria (Responders) compared to those subjects who did not meet the clinical stability criteria (Non-responders).
Mortality | 45 days
  Mortality rate at Day 45
Clinical Stability | 45 days
  Time (in days) to reach clinical stability (including survival status or excluding survival status)
Clinical Stability | 45 days
  Time (in days) to death
Clinical Stability | 45 days
  Time (in days) to hospital discharge of CS non-responders and death

CONTACTS AND LOCATIONS:
Locations (45):
- United States (45):
  - Mayo Clinic-Arizona, Phoenix, Arizona
  - City of Hope, Duarte, California
  - Children's Hospital of Orange County, Orange, California
  - Stanford University Medical Center, Palo Alto, California
  - UC Davis, Sacramento, California
  - Ansun Biopharma, Inc, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Lurie Children's Hospital, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Indiana Blood and Marrow Transplantation, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Children's Mercy Hospital, Kansas City, Kansas
  - University of Kansas, Kansas City, Kansas
  - John Hopkins University School of Medicine, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, School of Medicine, Minnesota City, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Weill Cornell Medical College/New York Presbyterian Hospital, New York, New York
  - Weill Cornell Medical College-Peds, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Stonybrook, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Nationwide Children's, Columbus, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt- Henry-Joyce Cancer Clinic, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Fred Hutchinson Cencer Research Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Chemaly RF, Marty FM, Wolfe CR, Lawrence SJ, Dadwal S, Soave R, Farthing J, Hawley S, Montanez P, Hwang J, Ho JH, Lewis S, Wang G, Boeckh M. DAS181 Treatment of Severe Lower Respiratory Tract Parainfluenza Virus Infection in Immunocompromised Patients: A Phase 2 Randomized, Placebo-Controlled Study. Clin Infect Dis. 2021 Aug 2;73(3):e773-e781. doi: 10.1093/cid/ciab113. PMID 33569576